CLINICAL TRIAL: NCT04144933
Title: A Randomized Control Trial Evaluating the Utility of Multimodal Opioid-free Anesthesia on Return of Bowel Function in Laparoscopic Colorectal Surgery
Brief Title: Effect of Multimodal Opioid-free Anesthesia on Return of Bowel Function in Laparoscopic Colorectal Surgery
Acronym: RUMBLE
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Saskatchewan (Other)
Responsible Party: Principal Investigator, Jonathan Gamble, Anesthesiologist, University of Saskatchewan
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: BIO-625
Record Dates: First submitted 2019-10-25; First posted 2019-10-30 (Actual); Last update posted 2023-12-20 (Actual); Status verified 2023-12

CONDITIONS: Anesthesia; General Anesthesia; Analgesics, Opioid; Opioid Free Anesthesia; Postoperative Ileus; Colorectal Surgery; Laparoscopic Surgery; Analgesia; Dexmedetomidine; Lidocaine; Ketamine
Keywords: Opioid-free; Opioid-sparing
MeSH Terms: conditions — Agnosia | interventions — Acetaminophen; Gabapentin; Lidocaine; Dexmedetomidine; Ketamine; Dexamethasone; Ondansetron; Sevoflurane; Magnesium Sulfate; Sufentanil

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Opioid-free General Anesthesia (OFA) (Experimental): Opioid-free preoperative medications, Opioid-free pre-intubation medications, Opioid-free maintenance medication, postoperative nausea and vomiting prophylaxis.
  Interventions: Drug: Acetaminophen, Gabapentin; Drug: Lidocaine 1% Injectable Solution, Dexmedetomidine, Ketamine; Drug: Dexamethasone, Ondansetron; Drug: Sevoflurane, Lidocaine 2% Injectable Solution, Ketamine, Dexmedetomidine, Magnesium Sulfate
- Traditional Opioid-containing General Anesthesia (TOA) (Active Comparator): Opioid-sparing preoperative medications, Opioid-containing pre-intubation medications, Opioid-containing maintenance medications, postoperative nausea and vomiting prophylaxis.
  Interventions: Drug: Acetaminophen, Gabapentin; Drug: Dexamethasone, Ondansetron; Drug: Lidocaine 1% Injectable Solution, Sufentanil; Drug: Sevoflurane, Sufentanil

INTERVENTIONS:
Drug: Acetaminophen, Gabapentin — 975 mg, 300 mg
  Other Names: Opioid-free preoperative medications
  Arms: Opioid-free General Anesthesia (OFA)
Drug: Acetaminophen, Gabapentin — 975 mg, 300 mg
  Other Names: Opioid-containing preoperative medications
  Arms: Traditional Opioid-containing General Anesthesia (TOA)
Drug: Lidocaine 1% Injectable Solution, Dexmedetomidine, Ketamine — 1.5 mg/kg, 0.5 mcg/kg, 0.5 mg/kg
  Other Names: Opioid-free pre-intubation medications
  Arms: Opioid-free General Anesthesia (OFA)
Drug: Dexamethasone, Ondansetron — 6 mg, 4 mg
  Other Names: Postoperative nausea and vomiting prophylaxis
Drug: Sevoflurane, Lidocaine 2% Injectable Solution, Ketamine, Dexmedetomidine, Magnesium Sulfate — Dose titrated to effect, 1.5 mg/kg/hr, 0.15 mg/kg/hr, 0.3 -1 mcg/kg/hr (titrated to effect), 30 mg/kg bolus over 30 minutes
  Other Names: Opioid-free maintenance medications
  Arms: Opioid-free General Anesthesia (OFA)
Drug: Lidocaine 1% Injectable Solution, Sufentanil — 0.5 mg/kg, 0.25-0.5 mcg/kg (titrated to effect)
  Other Names: Opioid-containing pre-intubation medications
  Arms: Traditional Opioid-containing General Anesthesia (TOA)
Drug: Sevoflurane, Sufentanil — Dose titrated to effect, As needed (dose at anesthesiologist's discretion)
  Other Names: Opioid-containing maintenance medications
  Arms: Traditional Opioid-containing General Anesthesia (TOA)

SUMMARY:
The objective of this study is to determine if an opioid-free general anesthetic (OFA) technique utilizing lidocaine, ketamine, dexmedetomidine and magnesium reduce postoperative opioid consumption and speed return of bowel function in patients undergoing elective, laparoscopic, colorectal surgery compared to traditional opioid-containing general anesthetic techniques. It is hypothesized that this intraoperative OFA regimen will reduce postoperative opioid consumption, and expedite return of bowel function in this population.

DETAILED DESCRIPTION:
The objective of this trial is to determine whether an opioid-free general anesthetic can help reduce postoperative opioid consumption and speed return of bowel function in patients undergoing elective, laparoscopic, colorectal surgery when compared with traditional opioid-containing techniques.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18, American Society of Anesthesiology (ASA) class I-III patients scheduled for elective laparoscopic/laparoscopic assisted colorectal surgery

Exclusion Criteria:

* Emergency surgery, open surgery, contraindications to laparoscopic surgery (ie. adhesions, inability to tolerate pneumoperitoneum), American Society of Anesthesiology (ASA) class 4, age < 18, pregnant or breastfeeding women, significant cardiorespiratory/hepatic/renal disease, allergy to any study drugs, inability to consent, inability to respond to pain assessments, inability to use the patient controlled analgesia device (PCA)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2021-05-15 (Actual); Primary Completion 2024-07-30 (Estimated); Study Completion 2024-08-01 (Estimated)

PRIMARY OUTCOMES:
Time to first flatus | End of surgery to first flatus (1-4 days)
  Time between the end of surgery and the movement when the patient first passes flatus

SECONDARY OUTCOMES:
Time to first defecation | End of surgery to first defecation (1-7 days)
  Time between the end of surgery and the moment the patient first passes stool
Time to tolerance of oral intake | End of surgery to first oral intake (1-3 days)
  Time between the end of surgery to when the patient can tolerate any oral solid food intake
Total Post-Anesthetic Care Unit (PACU) opioid consumption | End of surgery to discharge from PACU (1-2 hours)
  Total amount of opioid (morphine equivalents) required in PACU
Patient Controlled Analgesia (PCA) morphine consumption | End of surgery to 48 hours postoperatively
  Total amount of PCA morphine (mg) required from end of surgery to 48 hours postoperatively
Time to Post-Anesthetic Care Unit (PACU) discharge readiness | End of surgery to PACU discharge readiness (1-3 hours)
  Time to Post-Anesthetic Care Unit (PACU) discharge readiness
Visual Analogue Scale (VAS) pain scores | End of surgery to 48 hours postoperatively
  Visual Analogue Scale (VAS) pain scores will be recorded on a scale of 0 to 10, with 0 indicating no pain, and 10 indicating extreme pain, 48 hours following surgery
Quality of recovery after surgery | End of surgery to time of patient discharge from hospital (2-10 days)
  Assessed using the Quality of Recovery (QoR) 15 questionnaire, a validated tool for measuring quality of recovery after anesthesia and surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Royal University Hospital, Saskatoon, Saskatchewan, Canada

IPD SHARING:
Plan to Share IPD: No